CLINICAL TRIAL: NCT01867931
Title: Characterisation of Esophageal Epithelial Damage in Patients With Non-erosive Reflux Disease (NERD) and Erosive Esophagitis (EE): Role of Epithelial Permeability
Brief Title: Epithelial Damage in GERD
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL39721.068.12
Record Dates: First submitted 2013-04-04; First posted 2013-06-04 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Gastro-esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Erosive Esophagitis
- Non-erosive Reflux Disease
- Heatlhy volunteers

SUMMARY:
The purpose of this study is to characterize and compare epithelial damage in patients with erosive esophagitis and non-erosive reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Typical GERD-symptoms lasting for more than 6 months (recurrent episodes of heartburn or acid regurgitation)
* abnormal pH-parameters (pathological acid exposure and/or symptom association)

Exclusion Criteria:

* Age <18 years
* Previous esophageal or gastric surgery
* Severe esophageal motility disorder on manometry
* Histological evidence of Barrett's mucosa
* Severe co-morbidities (including cardiopulmonary disease, portal hypertension, collagen diseases, morbid obesity, coagulation disorders and co-morbidity hindering a gastroscopic procedure)
* Use of anticoagulant or immunosuppressive drugs
* Inability to stop medication that can influence the test results, like PPI, for at least 10 days before tests
* Excessive alcohol consumption (>20 units per week)
* Patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with EE and patients with NERD referred to the GI-outpatient clinic of the University Hospital Maastricht with an indication for diagnostic gastroscopy, as well healthy volunteers will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Epithelial integrity in tissue biopsies | 1 year

SECONDARY OUTCOMES:
Immunohistochemical markers in tissue biopsies | 1 year
Histological changes in tissue biopsies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: J.M. Conchillo, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Background] Jovov B, Que J, Tobey NA, Djukic Z, Hogan BL, Orlando RC. Role of E-cadherin in the pathogenesis of gastroesophageal reflux disease. Am J Gastroenterol. 2011 Jun;106(6):1039-47. doi: 10.1038/ajg.2011.102. Epub 2011 Mar 29. PMID 21448147
- [Background] Barlow WJ, Orlando RC. The pathogenesis of heartburn in nonerosive reflux disease: a unifying hypothesis. Gastroenterology. 2005 Mar;128(3):771-8. doi: 10.1053/j.gastro.2004.08.014. PMID 15765412